CLINICAL TRIAL: NCT02393625
Title: A Multi-center, Open-label Study to Assess the Safety and Efficacy of Combination Ceritinib (LDK378) and Nivolumab in Adult Patients With Anaplastic Lymphoma Kinase (ALK)-Positive Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study of Safety and Efficacy of Ceritinib in Combination With Nivolumab in Patients With ALK-positive Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2120C; 2024-510824-38-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2015-02-23; First posted 2015-03-19 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: ALK-positive NSCLC
Keywords: NSCLC, ALK-positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ceritinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental)
  Interventions: Drug: Ceritinib (LDK378); Drug: Nivolumab
- Dose Expansion (Experimental)
  Interventions: Drug: Ceritinib (LDK378); Drug: Nivolumab

INTERVENTIONS:
Drug: Ceritinib (LDK378)
Drug: Nivolumab

SUMMARY:
This is an open label multi center trial to determine the safety and efficacy of ceritinib in combination with nivolumab in ALK-positive NSCLC patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC that carries an ALK rearrangement
* Stage IIIB or IV NSCLC or relapsed locally advanced or metastatic NSCLC
* Presence of at least one measurable lesion as defined by RECIST 1.1
* Patients who have received prior chemotherapy, other ALK inhibitors, biologic therapy, or other investigational agents, must have recovered from all toxicities related to prior anticancer therapies to grade ≤1 (CTCAE v 4.03). Patients with grade ≤ 2 peripheral neuropathy or any grade of alopecia, fatigue, nail changes or skin changes are allowed to enter the study
* Patient has a WHO performance status 0-1

Exclusion Criteria:

* Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years
* Patients with an active, known or suspected autoimmune disease
* Unable or unwilling to swallow tablets or capsules
* Patient has other severe, acute, or chronic medical conditions including uncontrolled diabetes mellitus or psychiatric conditions or laboratory abnormalities that in the opinion of the Investigator may increase the risk associated with study participation, or that may interfere with the interpretation of study results

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Dose for Expansion | Study Day 42 (6 weeks)
Overall response rate (ORR) | 24 Weeks
  ORR (complete response (CR)+ partial response (PR)) per RECIST 1.1 as assessed by investigator

SECONDARY OUTCOMES:
Duration of Response (DOR) | 24 weeks
Disease Control Rate (DCR) | 24 weeks
Time to Response (TTR) | 24 weeks
Progression Free Survival (PFS) | 24 weeks
Overall survival (OS) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (4):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Thoracic Oncolgoy, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Novartis Investigative Site, Heidelberg, Victoria, Australia
- Novartis Investigative Site, Leuven, Vlaams Brabant, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spigel DR, Reynolds C, Waterhouse D, Garon EB, Chandler J, Babu S, Thurmes P, Spira A, Jotte R, Zhu J, Lin WH, Blumenschein G Jr. Phase 1/2 Study of the Safety and Tolerability of Nivolumab Plus Crizotinib for the First-Line Treatment of Anaplastic Lymphoma Kinase Translocation - Positive Advanced Non-Small Cell Lung Cancer (CheckMate 370). J Thorac Oncol. 2018 May;13(5):682-688. doi: 10.1016/j.jtho.2018.02.022. Epub 2018 Mar 6. PMID 29518553